CLINICAL TRIAL: NCT03242707
Title: A Randomized, Controlled Study to Evaluate the Efficacy of Intra-articular, Autologous Adipose Tissue Injections for the Treatment of Mild-to-Moderate Osteoarthritis
Brief Title: Intra-articular Adipose Tissue Injections for Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Thomas Vangsness, Professor of Orthopaedic Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-17-00365
Record Dates: First submitted 2017-07-28; First posted 2017-08-08 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either a single autologous fat injection or a single hyaluronic acid injection.
Masking Description: Patients will know which group they have been assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous adipose tissue knee injection (Experimental): Fat will be removed from the abdomen and processed using the Lipogems device. Approximately 5ml of the microfragmented fat product will be injected into the knee joint.
  Interventions: Biological: Autologous adipose tissue injection
- Hyaluronic Acid knee injection (Active Comparator): Hyaluronic Acid - Synvisc-One®: A high molecular weight sodium hyaluronate (HA). HA is an FDA approved, standard of care treatment.
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Biological: Autologous adipose tissue injection — 20ml to 40ml of subcutaneous adipose tissue will be aspirated from the abdomen. Adipose tissue will be processed using the Lipogems device, a closed-loop processing device used in medical procedures involving the harvesting, concentrating and transferring of autologous adipose tissue.
  The resulting fat product will be delivered locally via ultrasound-guided, intra-articular injection.
  Other Names: Lipogems, Microfragmented fat
  Arms: Autologous adipose tissue knee injection
Drug: Hyaluronic Acid — Synvisc-One® is a high molecular weight sodium hyaluronate.
  Arms: Hyaluronic Acid knee injection

SUMMARY:
A new generation of "minimally manipulated" regenerative treatments are being offered at clinics across the country, but there is no strong efficacy data to support their use. The purpose of this study is to estimate the effect size of the treatment by comparing the efficacy of autologous fat to the current standard of care treatment, hyaluronic acid (HA). As a secondary aim, we will test for preliminary evidence of efficacy of autologous fat vs. HA and determine how these treatments effect the biochemical environment of the knee by comparing pre-injection and post-injection synovial fluid biomarker profiles.

DETAILED DESCRIPTION:
In recent years, fat treatments administered for structural reconstruction, repair, or replacement are being increasingly offered at clinics across the country. These treatments contain both autologous cells that are often referred to as "stem cells" or "MSCs" and extra-cellular matrix (ECM). Cell therapies containing ECM are thought to have the following advantages over treatments prepared using enzymatic digestion: (1) preservation of the stromal vascular niche, which allows time-release of the regenerative factors; (2) release of bioactive molecules by exosomes, which have been demonstrated to be significantly greater in mechanically processed fat than enzymatically processed fat; and (3) maintenance of the structural and morphologic unit, which is thought to increase cell efficacy by making the cells more resilient to the harsh conditions in the recipient environment. Case reports investigating the use of autologous fat treatments show promise, but a number of questions remain unanswered. Agents injected into the joint tend to be quickly cleared from the body and ECM itself has the potential to produce inflammatory signals and induce osteoarthritis.

This study will use a Hyaluronic acid (HA) as an active control, which is the standard of care for pain associated with osteoarthritis. The use of HA as an active control for autologous cell-based therapies is well established and is the best option given the need to aspirate fat tissue from patients who will be receiving the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 to 75, inclusive
2. Normal axial alignment
3. X-ray, Kellgren-Lawrence OA grade 2 - 3, inclusive
4. WOMAC-pain: Between 9 and 19, inclusive
5. Willingness to participate all scheduled follow-ups
6. Willingness to refrain from taking NSAIDs, level 2 analgesics, and opioids for the course of the study
7. BMI < 40

Exclusion Criteria:

1. Pregnant or lactating
2. Intra-articular injection within 3 months of treatment
3. Inflammatory arthritis
4. Any disease or active drug use that significantly compromises coagulation
5. Significant damage and/or tears of the ACL or other supporting tissues
6. Prior knee surgery in the last 6 months in the knee that will be injected
7. Active tobacco use
8. Active alcohol or substance abuse within 6 months of study entry
9. Known hypersensitivity (allergy) to hyaluronan (sodium hyaluronate) preparations
10. Knee joint infections, skin diseases or infections in the area of the injection site
11. Diabetes
12. Active inhaler use
13. Any medical condition, which in the opinion of the clinical investigator, would interfere with the treatment or outcome evaluation

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The pain items of then Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC-A) | Change from baseline WOMAC score at 6 months
  WOMAC-A is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System 29-item (PROMIS®-29) | Change from baseline in PROMIS-29 from baseline to 6 months
  A collection of 4-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Western Ontario and McMaster Universities Osteoarthritis Index | Change from baseline in PROMIS-29 from baseline to 6 months
  WOMAC is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
Clinical Anchors | Clinical anchors from baseline to 6 months
  Clinical anchors will be used to identify minimal important differences in treatment groups

OTHER OUTCOMES:
Synovial fluid analysis | Baseline, 6 weeks and 6 months
  Selected OA biomarker profiles that define different OA phenotypes predict the responses to autologous adipose tissue injections
Short-term clinical evaluation - WOMAC | Change from baseline at 6 weeks
  WOMAC questionnaire will be administered at the 6-week follow-up
Short-term clinical evaluation - PROMIS | Change from baseline at 6 weeks
  PROMIS questionnaire will be administered at the 6-week follow-up
Force Plate Analysis | Assessment and change from baseline to 6 weeks and 6 months
  Balance will be assessed using a proprietary force plate system at baseline, 6 weeks and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: C.Thomas Vangsness, MD, Principal Investigator — Keck School of Medicine of USC
Locations (1):
- Keck Medicine of USC, Los Angeles, California, United States

REFERENCES:
- [Derived] Jones IA, Wilson M, Togashi R, Han B, Mircheff AK, Thomas Vangsness C Jr. A randomized, controlled study to evaluate the efficacy of intra-articular, autologous adipose tissue injections for the treatment of mild-to-moderate knee osteoarthritis compared to hyaluronic acid: a study protocol. BMC Musculoskelet Disord. 2018 Oct 24;19(1):383. doi: 10.1186/s12891-018-2300-7. PMID 30355323